CLINICAL TRIAL: NCT01683201
Title: Functional Exercise After Total Hip Replacement: A Randomised Controlled Late Phase Trial
Brief Title: Functional Exercise After Total Hip Replacement
Acronym: FEATHER
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Health Service Executive, Ireland (Other)
Responsible Party: Principal Investigator, Brenda Monaghan, Principal Investigator Clinical Specialist Physiotherapist, Health Service Executive, Ireland
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: HPF/2011/60
Record Dates: First submitted 2012-09-07; First posted 2012-09-11 (Estimated); Last update posted 2015-03-20 (Estimated); Status verified 2015-03

CONDITIONS: Hip Surgery Corrective
Keywords: Total hip replacement; Functional exercise class; Randomised controlled trial

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Functional exercise class (Experimental): Functional exercise class 45 mins twice weekly from week 12 to week 18
  Interventions: Procedure: Functional exercise class
- Usual Care Group (Placebo Comparator): Usual Care
  Interventions: Procedure: usual care group

INTERVENTIONS:
Procedure: Functional exercise class — Functional exercise class running twice weekly for six weeks from week 12 to week 18
  Arms: Functional exercise class
Procedure: usual care group — Usual care group adhere to post operative instructions given on discharge from hospital
  Arms: Usual Care Group

SUMMARY:
The aim of this research project is to evaluate the efficacy of a specific functional exercise programme to improve pain, stiffness and physical function in patients post total hip replacement from week 12 to week 18 post surgery.

DETAILED DESCRIPTION:
This will be a single blind randomised controlled trial with two arms. 70 subjects post primary total hip replacement will be randomised either to a functional; exercise group (n=35) or to a control group following usual care (n=35).

Blinded outcome assessments will be carried out on all subjects by the principal investigator using the Western Ontario and Mc Master arthritis index on day 5 , week 12 aand week 18.

Secondary outcomes measurements will also be collated at week 12 and week 18 including SF 12, 6 min walk test, Dynamometry, and a blinded radiologist will also measure glut med cross sectional area using real time ultrasound at week 12 and week 18.

ELIGIBILITY:
Inclusion Criteria:

* 12 weeks post primary THR for osteoarthritis
* Age 50 years and above
* Able to read and understand and instructions in English
* Willing to attend classes twice weekly for 8 weeks
* Able to participate in an exercise programme without physical assistance
* Able to Mobilize independently 15m without crutches and /or stick -Passed by the referring Orthopaedic Consultant as suitable for inclusion at six week appointment -

Exclusion Criteria:

* Medically unstable
* Any central or peripheral nervous system deficits
* Any underlying terminal disease -Any suspicion of infection following joint replacement -

Min Age: 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 72 (Actual)
Dates: Start 2012-09; Primary Completion 2014-01 (Actual); Study Completion 2015-02 (Actual)

PRIMARY OUTCOMES:
WOMAC Western Ontario and Mc Master osteoarthritis index questionaire | 3 YEARS
  Multi dimensional self administered health status instrument used to measure changes in the dimensions of pain stiffness and function.

SECONDARY OUTCOMES:
Six minute walk test, | 3 years
  Physical performance test used to measure the distance covered in a set timeframe.
Short form SF- 12 | 3 YEARS
  Self completed questionaire that measures health status and quality of life under eight multi item scales measuring physical function, bodily pain, role limitation due to physical health problems, general health, vitality, social function, role limitation due to emotional problems and mental health.
HiP Abduction Strength Dynamometry | 3 years
  Assessment scale of ability to maintain balance both statically and whilst performing various functional tasks will be completed by the principal investigator at week 12 and repeated for all patients at week 18.
Real time ultrasound imaging of the gluteus medius muscles | 3 years
  Patients will be scanned by a blinded radiologist to measure cross sectional area of the gluteus medius muscle at 12 weeks and again at 18 weeks.

CONTACTS AND LOCATIONS:
Overall Officials: Brenda M Monaghan, BSc, MSc, Principal Investigator — HSE Ireland

REFERENCES:
- [Derived] Monaghan B, Cunningham P, Harrington P, Hing W, Blake C, O' Dohertya D, Cusack T. Randomised controlled trial to evaluate a physiotherapy-led functional exercise programme after total hip replacement. Physiotherapy. 2017 Sep;103(3):283-288. doi: 10.1016/j.physio.2016.01.003. Epub 2016 Feb 15. PMID 27126617
- [Derived] Monaghan B, Grant T, Hing W, Cusack T. Functional exercise after total hip replacement (FEATHER): a randomised control trial. BMC Musculoskelet Disord. 2012 Nov 28;13:237. doi: 10.1186/1471-2474-13-237. PMID 23190932